CLINICAL TRIAL: NCT00005208
Title: Regulation of Placental Vascular Reactivity in Pregnancy-induced Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1087; R01HL040029 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Pregnancy Toxemias
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Pre-Eclampsia

SUMMARY:
To elucidate the role of an imbalance in vasodilator prostacyclin (PGI2) and vasoconstrictor thromboxane (TxA2) in pregnancy-induced hypertension

DETAILED DESCRIPTION:
BACKGROUND:

Pregnancy-induced hypertension (PIH) is associated with increased fetal and neonatal morbidity and mortality possibly resulting from hypoxia in utero. The primary pathology of PIH involves a reduction in uteroplacental blood flow but modern imaging techniques have now shown that increased impedance of the fetal-placental circulation and hence reduced blood flow can also be found in PIH. This may represent a direct effect of hypoxia or be a fetal adaptation to increase placental oxygen extraction to relieve hypoxia. The fetal-placental circulation is regulated by humoral agents and vascular pressure. An imbalance of vasodilator prostacyclin (PGI2) and vasoconstrictor thromboxane (TxA2) production is reported to underlie the vasoconstriction seen in PIH.

The study resulted from the 1986 release of a Request for Applications for Research on Hypertension in Pregnancy by the National Heart, Lung, and Blood Institute and the National Institute of Child Health and Human Development.

DESIGN NARRATIVE:

The fetal-placental circulations of perfused human placental cotyledons from normotensive and pregnancy-induced hypertensive pregnancies were used to determine if an imbalance in PGI2/TxA2 production existed and its relationship to the responses of the fetal-placental circulation to vasoconstriction. Studies were also conducted on the effects of hypocalcemia and hypomagnesemia, hypoxia, and drugs.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1987-09; Study Completion 1992-07 (Actual)

REFERENCES:
- [Background] Myatt L, Brewer AS, Brockman DE. The comparative effects of big endothelin-1, endothelin-1, and endothelin-3 in the human fetal-placental circulation. Am J Obstet Gynecol. 1992 Dec;167(6):1651-6. doi: 10.1016/0002-9378(92)91756-z. PMID 1471681
- [Background] Myatt L. Control of vascular resistance in the human placenta. Placenta. 1992 Jul-Aug;13(4):329-41. doi: 10.1016/0143-4004(92)90057-z. No abstract available. PMID 1438081
- [Background] Eis AW, Mitchell MD, Myatt L. Endothelin transfer and endothelin effects on water transfer in human fetal membranes. Obstet Gynecol. 1992 Mar;79(3):411-5. doi: 10.1097/00006250-199203000-00017. PMID 1738524
- [Background] Myatt L, Brewer AS, Langdon G, Brockman DE. Attenuation of the vasoconstrictor effects of thromboxane and endothelin by nitric oxide in the human fetal-placental circulation. Am J Obstet Gynecol. 1992 Jan;166(1 Pt 1):224-30. doi: 10.1016/0002-9378(92)91863-6. PMID 1733199
- [Background] Myatt L, Langdon G, Brewer AS, Brockman DE. Endothelin-1-induced vasoconstriction is not mediated by thromboxane release and action in the human fetal-placental circulation. Am J Obstet Gynecol. 1991 Dec;165(6 Pt 1):1717-22. doi: 10.1016/0002-9378(91)90021-i. PMID 1750466
- [Background] Jacobson RL, Brewer A, Eis A, Siddiqi TA, Myatt L. Transfer of aspirin across the perfused human placental cotyledon. Am J Obstet Gynecol. 1991 Oct;165(4 Pt 1):939-44. doi: 10.1016/0002-9378(91)90444-v. PMID 1951559
- [Background] Myatt L, Brewer A, Brockman DE. The action of nitric oxide in the perfused human fetal-placental circulation. Am J Obstet Gynecol. 1991 Feb;164(2):687-92. doi: 10.1016/s0002-9378(11)80047-5. PMID 1899534
- [Background] Myatt L, Brockman DE, Langdon G, Pollock JS. Constitutive calcium-dependent isoform of nitric oxide synthase in the human placental villous vascular tree. Placenta. 1993 Jul-Aug;14(4):373-83. doi: 10.1016/s0143-4004(05)80459-x. PMID 7504255